CLINICAL TRIAL: NCT00252824
Title: A Comparison of the Efficacy of Symbicort® Single Inhaler Therapy (Symbicort Turbuhaler® 160/4.5 mg 1 Inhalation b.i.d. Plus As-needed) and Conventional Best Practice for the Treatment of Persistent Asthma in Adolescents and Adults - a 26 Weeks, Randomised, Open-label, Parallel-group, Multicentre Study
Brief Title: STYLE - Symbicort Single Inhaler Therapy vs Conventional Therapy in Treatment of Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00014; STYLE
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: Budesonide/formoterol Turbuhaler vs Conventional Best Asthma Therapy
  Other Names: Symbicort

SUMMARY:
The purpose of the study is to compare the efficacy of a flexible dose of Symbicort with conventional stepwise treatment according to asthma treatment guidelines in patients with persistent asthma

ELIGIBILITY:
Inclusion Criteria:

* - Diagnosis of asthma ³ 3 months
* Prescribed daily use of glucocorticosteroids at a dose > 320 mcg/ day for at least 3 months prior to Visit 1

Exclusion Criteria:

* Smoking history > 10 pack-years
* Asthma exacerbation requiring change in asthma treatment during the last 14 days prior to inclusion
* Any significant disease or disorder that my jeopardize the safety of the patient.

Additional inclusion and exclusion criteria will be evaluated by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2005-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Time to first severe asthma exacerbation

SECONDARY OUTCOMES:
Number of asthma exacerbations
Mean use of as-needed medication
Prescribed asthma medication
Asthma Control Questionnaire
Asthma related costs (direct asthma medication, direct non-medication costs and indirect costs)
Safety: Serious Adverse Events and discontinuations due to adverse events
All variables assessed over the 6 months treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (53):
- Chile (2):
  - Research Site, Quillota
  - Research Site, Valparaíso
- Croatia (3):
  - Researh Site, Dubrovnik
  - Research Site, Split
  - Research Site, Zagreb
- Czechia (8):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Litomice
  - Research Site, Ostrava
  - Research Site, Prague
  - Research Site, Prostijov
  - Research Site, Strakonice
- Greece (4):
  - Research Site, Ahens
  - Research Site, Alexandroup
  - Research Site, Athens
  - Research Site, Kavala
- Iceland (2):
  - Research Site, Akureyri
  - Research Site, Reykjavik
- Latvia (3):
  - Research Site, Daugavpils
  - Research Site, Riga
  - Research Site, Rigas Raj
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Portugal (7):
  - Research Site, Aveiro
  - Research Site, Coimbra
  - Research Site, Coviha
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Setúbal
  - Research Site, Vila Nova de Gaia
- Slovakia (13):
  - Research Site, Banská Bystrica
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Hlohovec
  - Research Site, Košice
  - Research Site, Liptovský Hrádok
  - Research Site, Malacky
  - Research Site, Nitra Zobor
  - Research Site, Partizánske
  - Research Site, Revúca
  - Research Site, Senec
  - Research Site, Topostany
  - Research Site, Žilina
- Slovenia (8):
  - Research Site, Celje
  - Research Site, Golnik
  - Research Site, Kamnik
  - Research Site, Koper
  - Research Site, Litija
  - Research Site, Ljubljana
  - Research Site, Murska Sobota
  - Research Site, Nova Gorica